CLINICAL TRIAL: NCT04807816
Title: Targeting ATR in Soft-tissue Sarcomas: a Randomized Phase II Study. TARSARC Study
Brief Title: Targeting ATR in Soft-tissue Sarcomas
Acronym: TARSARC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IB 2018-04; 2018-003835-31 (EudraCT Number)
Record Dates: First submitted 2021-03-15; First posted 2021-03-19 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Leiomyosarcoma, Adult
Keywords: ATR inhibition; soft-tissue sarcoma; advanced/metastatic
MeSH Terms: conditions — Leiomyosarcoma; Sarcoma; Neoplasm Metastasis | interventions — Gemcitabine

STUDY DESIGN:
Intervention Model Description: This is a multicenter, prospective, open-labeled, 2-arm, non-comparative randomized (2:1) phase II trial. Patients will be randomized between arm A (gemcitabine + berzosertib) and arm B (gemcitabine) with two patients randomized in arm A for one patient randomized in arm B.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm A: treatment by berzosertib combined with gemcitabine (Experimental): Patients with advanced leiomyosarcomas will be treated with berzosertib combined with gemcitabine
  Interventions: Drug: Association of berzosertib with gemcitabine
- Standard Arm B: treatment by gemcitabine alone (Other): Patients with advanced leiomyosarcomas will be treated with with gemcitabine alone (control arm)
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Association of berzosertib with gemcitabine — Gemcitabine will be administered by intravenous 30-minutes infusion on days 1 and 8 every 3 weeks, at a fixed dose of 1000 mg/m².
  Berzosertib will be administered intravenously on days 2 and 9 every 3 weeks (210 mg/m²).
  A treatment cycle consists of 3 weeks (i.e., 21 days) and will be administered during hospitalization.
  Other Names: Experimental
  Arms: Experimental Arm A: treatment by berzosertib combined with gemcitabine
Drug: Gemcitabine — Gemcitabine will be administered by intravenous 30-minutes infusion on days 1 and 8 every 3 weeks, at a fixed dose of 1000 mg/m².
  A treatment cycle consists of 3 weeks (i.e., 21 days) and will be administered during hospitalization.
  Other Names: Control
  Arms: Standard Arm B: treatment by gemcitabine alone

SUMMARY:
Multicenter, prospective, open-labeled, 2-arm, non-comparative randomized phase II trial to assess the antitumor activity of berzosertib in association with gemcitabine

DETAILED DESCRIPTION:
This is a multicenter, prospective, open-labeled, 2-arm, non-comparative randomized (2:1) phase II trial. Patients will be randomized between arm A (gemcitabine + berzosertib) and arm B (gemcitabine) with two patients randomized in arm A for one patient randomized in arm B.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed leiomyosarcomas.
2. Metastatic or unresectable locally advanced disease,
3. Documented progression according to RECIST v1.1 confirmed by central review,
4. Age ≥ 18 years,
5. ECOG ≤ 1,
6. Life expectancy > 3 months,
7. No more than 3 previous line of systemic therapy for advanced disease,
8. Patients must have advanced disease and must not be a candidate for other approved therapeutic regimen known to provide significant clinical benefit based on investigator judgement,
9. Patients must have measurable disease defined as per RECIST v1.1
10. Patient must comply with the collection of tumor biopsies, and tumors must be accessible for biopsy,
11. At least three weeks since last chemotherapy, immunotherapy or any other pharmacological treatment and/or radiotherapy,
12. Adequate hematological, renal, metabolic and hepatic function
13. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to randomization.
14. Both women of childbearing potential and men must agree to use a highly effective method of contraception 28 days before start of first dose of study drug
15. No prior or concurrent malignant disease diagnosed or treated in the last 2 years except for adequately treated in situ carcinoma of the cervix, basal or squamous skin cell carcinoma, or in situ transitional bladder cell carcinoma,
16. Recovery to grade ≤ 1 from any adverse event (AE) derived from previous treatment
17. Voluntarily signed and dated written informed consent prior to any study specific procedure,
18. Patients with a social security in compliance with the French law.

Exclusion Criteria:

1. Previous treatment with Gemcitabine, or berzosertib or other ATR inhibitor,
2. Evidence of progressive or symptomatic central nervous system or leptomeningeal metastases,
3. Women who are pregnant or breast feeding,
4. Participation to a study involving a medical or therapeutic intervention in the last 30 days,
5. Previous enrolment in the present study,
6. Patient unable to follow and comply with the study procedures because of any geographical, social or psychological reasons,
7. Known hypersensitivity to any involved study drug or any of its formulation components,
8. Has known active hepatitis B or hepatitis C,
9. Has a known history of Human Immunodeficiency Virus or known acquired immunodeficiency syndrome
10. Any of the following cardiac or cardiovascular criteria :

    * Congestive heart failure ≥ New York Heart Association (NHYA) class 1,
    * Unstable angina , new-onset angina
    * Myocardial infarction less than 6 months before start of study drug
    * Uncontrolled cardiac arrhythmias,
11. Participants with Li Fraumeni syndrome and/or ataxia telangiectasia,
12. Active autoimmune disease:

    * Patients with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible,
    * Patients requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at dose ≤ 10 mg or 10 mg equivalent prednisone day,
    * Administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intra-ocular or inhalation) are acceptable.
13. Arterial or venous thrombotic or embolic events such as cerebrovascular accident , deep vein thrombosis or pulmonary embolism within 6 months before the start of study medication,
14. Patients with oral anticoagulation based on Vitamine K antagonist,
15. Treatment by potent inhibitors or inducers of CYP3A4
16. Vaccination with yellow fever or by any other live attenuated vaccine in the last 30 days,
17. Individuals deprived of liberty or placed under legual guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-02-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of the antitumor activity of berzosertib combined with gemcitabine | 6 months
  Antitumor activity will be assessed in terms of 6-month progression-free rate and is defined as the rate of complete or partial response (CR, PR) or stable disease (SD), as per RECIST v1.1.
Assessment of the antitumor activity of gemcitabine | 6 months
  Antitumor activity will be assessed in terms of 6-month progression-free rate and is defined as the rate of complete or partial response (CR, PR) or stable disease (SD), as per RECIST v1.1.

SECONDARY OUTCOMES:
6-month objective response rate (ORR) for patients treated by berzosertib in association with gemcitabine | 6 months
  Objective response is defined as complete response (CR) or partial response (PR) as per adapted RECIST v1.1.
6-month objective response rate (ORR) for patients treated by gemcitabine alone | 6 months
  Objective response is defined as complete response (CR) or partial response (PR) as per adapted RECIST v1.1.
Best overall response for patients treated by berzosertib in association with gemcitabine | throughout the treatment period, an expected average of 6 months
  Best overall response is defined as the best reponse across all time points (RECIST v1.1). The best overall response rate is determined once all the data for the patient is known
Best overall response for patients treated by gemcitabine alone | throughout the treatment period, an expected average of 6 months
  Best overall response is defined as the best reponse across all time points (RECIST v1.1). The best overall response rate is determined once all the data for the patient is known
1-year progression-free survival for patients treated by berzosertib in association with gemcitabine | 1 year
  Progression-free survival is defined as the delay between the start date of treatment and the date of progression (as per RECIST v1.1) or death (from any cause), whichever occurs first
1-year progression-free survival for patients treated by gemcitabine alone | 1 year
  Progression-free survival is defined as the delay between the start date of treatment and the date of progression (as per RECIST v1.1) or death (from any cause), whichever occurs first
2-year progression-free survival for patients treated by berzosertib in association with gemcitabine | 2 years
  Progression-free survival is defined as the delay between the start date of treatment and the date of progression (as per RECIST v1.1) or death (from any cause), whichever occurs first
2-year progression-free survival for patients treated by gemcitabine alone | 2 years
  Progression-free survival is defined as the delay between the start date of treatment and the date of progression (as per RECIST v1.1) or death (from any cause), whichever occurs first
1-year overall survival for patients treated by berzosertib in association with gemcitabine | 1 year
  Overall survival is defined as the delay between the start date of treatment and the date of death (from any cause)
1-year overall survival for patients treated by gemcitabine alone | 1 year
  Overall survival is defined as the delay between the start date of treatment and the date of death (from any cause)
2-year overall survival for patients treated by berzosertib in association with gemcitabine | 2 years
  Overall survival is defined as the delay between the start date of treatment and the date of death (from any cause)
2-year overall survival for patients treated by gemcitabine alone | 2 years
  Overall survival is defined as the delay between the start date of treatment and the date of death (from any cause)
6-month objective response according to CHOI criteria, independently for each arm | 6 months
  Objective response is defined as complete response (CR) or partial response (PR) as per CHOI criteria.
Best overall response according to CHOI criteria, independently for each arm | throughout the treatment period, an expected average of 6 months
  Best overall response is defined as the best reponse across all time points (CHOI criteria). The best overall response rate is determined once all the data for the patient is known
Safety profile independently for each arm: Common Terminology Criteria for Adverse Event version 5 | throughout the treatment period, an expected average of 6 months
  Toxicity graded using the Common Terminology Criteria for Adverse Events version 5
Tumor immune cells levels | before treatment onset and cycle 2 day 1 (each cycle is 21 days)
  Levels of immune cells (CD4, CD8, PDL1)in tumor will be measured by immunohistochemistry
Blood cytokines levels | baseline, cycle 2 day 1, cycle 6 day 1 and progression (each cycle is 21 days)
  Levels of cytokines (tryptophane, interleukine) in blood will be measured by ELISA
Blood lymphocytes levels | baseline, cycle 2 day 1, cycle 6 day 1 and progression (each cycle is 21 days)
  Levels of fixed PBMC (peripheral blood mononucear cells) in blood will be measured by flow cytometry
Blood kynurenine levels | baseline, cycle 2 day 1, cycle 6 day 1 and progression (each cycle is 21 days)
  Levels of kynurenine in blood will be measured by ELISA

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Institut Bergonié, Bordeaux
  - Centre Leon Berard, Lyon
  - CHU Poitiers, Poitiers
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - IUCT Oncopôle, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No